CLINICAL TRIAL: NCT02794922
Title: Effectiveness of Vitamin B in Reducing Temporomandibular Joint Disorder Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Winnie W.S. Choi, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW 15 - 266
Record Dates: First submitted 2016-05-30; First posted 2016-06-09 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Temporomandibular Joint Disorder
Keywords: Vitamin B; Temporomandibular joint disorder; trpv1
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Vitamin B Complex; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Interventional (Experimental): Name: Neurovit Forte tab Dosage: Each tablet contains Vitamin B1 242.5mg, Vitamin B6 250mg, Vitamin B12 1mg Frequency: One tab, once per day Duration: 6 weeks
  Interventions: Drug: Neurovit Forte
- Placebo (Placebo Comparator): Capsule containing 250mg corn starch
  Interventions: Drug: Corn Starch

INTERVENTIONS:
Drug: Neurovit Forte
  Other Names: Vitamin B Complex
  Arms: Interventional
Drug: Corn Starch
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine effectiveness of vitamin B in reducing temporomandibular joint disorder (TMD) pain. Patients will be randomised to receive the study drug or placebo. The study drug we are using is a combination of vitamin B1(thiamine mononitrate)-242.5mg; vitamin B6(pyridoxineHCl)-250mg, and vitamin B12(cyanocobalamin)-1mg. We will assess patient's pain level, range of jaw movement and record any side effects from using this medication.

DETAILED DESCRIPTION:
Type of study : Prospective double blinded randomized control trial Sample population : patients with temporomandibular joint disorder pain who are currently undergoing treatment in Oral & Maxillofacial surgery unit, Prince Philip Dental Hospital Study Period : 2 year (1st may2015 to 1st may 2017)

Data Collection All new cases or existing TMD patients treated in oral maxillofacial surgery department, Prince Philip Dental Hospital will be acquired and screened based on inclusion and exclusion criteria. Selected patients will be categorised based on TMD axis 1 diagnosis and divided into two groups - group 1(Vitamin B) and group 2(placebo) randomly . Allocation of patients into the group will be based on computer generated by random block sequence.

Complete social demographic background of the patient will recorded according to the following format age, gender, race, education, and job.

Clinical assessment will be done to check 1. Mouth opening 2. Lateral excursion (right and left) 3. Protrusion 4. Deviation of lower jaw on opening 5. Tenderness of muscle of mastication 6. Pain - based on 10cm visual analog score.

After initial assessments, patients will be started on either vitamin B complex or placebo based on their group.

* Both group of patients will be also prescribed with Tab Ibuprofen 400mg to be taken during acute Temporomandibular joint (TMJ) pain symptoms.
* These patients will be reviewed on week 0,2,4 and 6.
* All the patients will be reviewed by blinded assessor. Each patient will be given a log book to document frequency of TMJ pain attack, maximum pain score on each attack and amount of analgesics (Ibuprofen 400mg tabs) taken.
* Log book record will be checked on their review.
* Amount of analgesics recorded in log book and compliance of Vitamin B or placebo will be cross checked with remaining tablet count.

Data Evaluation/ Statistical Analyses The statistical analysis of this study will use the standard version of Statistical Package for the Social Sciences (SPSS) version 17.0 for windows. All the data will be gathered and entered in into this software.

ELIGIBILITY:
Inclusion Criteria:

* minimum age of 18
* temporomandibular joint disorder with pain
* chronic condition- symptoms lasting more than 3 months with at least 2 episodes of pain in last 1 month
* language competence- in Cantonese or English
* all ethnicity

Exclusion Criteria:

* ankylosis of the joint
* limited mental capacity
* pregnancy and lactating mothers
* inability to take medications (NSAIDS-Ibuprofen or Vitamin B)
* undergoing concurrent pharmacotherapy with anti inflammatory or muscle relaxant medications
* poor general health
* history of TMJ trauma or TMJ surgery
* subjects taking Vitamin B for other uses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale(VAS) Pain Score | baseline
  assessment of pain level with VAS score at baseline (week 0)
Visual Analog Scale(VAS) Pain Score | week 2
  assessment of pain level with VAS score at week2
Visual Analog Scale(VAS) Pain Score | week 4
  assessment of pain level with VAS score at week4
Visual Analog Scale(VAS) Pain Score | week 6
  assessment of pain level with VAS score at week6

SECONDARY OUTCOMES:
mouth opening measurement in millimeter (mm) | baseline
  assessment of mouth opening in millimeter (mm) at baseline (week0)
mouth opening measurement in millimeter (mm) | week 2
  assessment of mouth opening in millimeter (mm) at week 2
mouth opening measurement in millimeter (mm) | week4
  assessment of mouth opening in millimeter (mm) at week 4
mouth opening measurement in millimeter (mm) | week 6
  assessment of mouth opening in millimeter (mm) at week 6
number of participants with treatment related adverse events as assessed by CTCAE v4.03 | 6 weeks
  Subjects will be assessed for any adverse events related to intervention , by using CYCAE v4.03, at week 0, week 2, week 4 and week 6
tablet count measurements to check complaince | 6 weeks
  remaining tablets will be counted at end of Week 6 to check compliance rate towards treatment

CONTACTS AND LOCATIONS:
Overall Officials: Winnie Wing Shan Choi, BDS, MDS, Study Director — Faculty of Dentistry, The University of Hong Kong; Jothi R Rajaran, DDS, Principal Investigator — Faculty of Dentistry, The University of Hong Kong
Locations (1):
- Prince Philip Dental Hospital, Hong Kong, China